CLINICAL TRIAL: NCT03217084
Title: Esthetic Effect of Casein Phosphopeptide-Amorphous Calcium Phosphate Varnish Versus Tricalcium Phosphate Varnish on Postorthodontic White Spot Lesions: A Randomized Pilot Study
Brief Title: Treatment of Postorthodontic White Spot Lesions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelrahman Yousef ALduqi, Master degree student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FODM CU
Record Dates: First submitted 2017-07-12; First posted 2017-07-13 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: White Spot Lesion of Tooth
Keywords: White spot lesion ,fluoride varnish

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MI varnish GC (Active Comparator): MI Varnish is a 5% sodium fluoride varnish that has a desensitizing action when applied to tooth surfaces. MI Varnish also contains RECALDEN Open the unit-dose package of Varnish. Use the applicator brush to thoroughly mix Varnish . Apply Varnish evenly in a thin layer over treatment area(s). For larger surface areas, apply Varnish in sweeping horizontal brush. After application, instruct the patient to close his or her mouth to set the Varnish. No need to use suction. The patient may feel the thin coating when rubbing the treated area with his or her tongue.
  Interventions: Drug: MI varnish GC
- White Varnish 3M (Active Comparator): White Varnish is a 5% sodium fluoride varnish that has a desensitizing action when applied to tooth surfaces. White Varnish an innovative tri-calcium phosphate.
  Open the unit-dose package of Varnish. Use the applicator brush to thoroughly mix Varnish . Apply Varnish evenly in a thin layer over treatment area(s). For larger surface areas, apply Varnish in sweeping horizontal brush. After application, instruct the patient to close his or her mouth to set the Varnish. No need to use suction. The patient may feel the thin coating when rubbing the treated area with his or her tongue.
  Interventions: Drug: White varnish 3M

INTERVENTIONS:
Drug: MI varnish GC — MI Varnish GC is a 5% sodium fluoride varnish that has a desensitizing action when applied to tooth surfaces. MI Varnish also contains RECALDENT. Open the unit-dose package of Varnish. Use the applicator brush to thoroughly mix Varnish. Apply Varnish evenly in a thin layer over treatment area(s). For larger surface areas, apply Varnish in sweeping horizontal brush. After application, instruct the patient to close his or her mouth to set the Varnish. No need to use suction. The patient may feel the thin coating when rubbing the treated area with his or her tongue. The treatment period for Varnish is minimally 4 hour.
  Other Names: Fluoride Varnish
  Arms: MI varnish GC
Drug: White varnish 3M — White varnish 3M is a 5% sodium fluoride varnish that has a desensitizing action when applied to tooth surfaces. Clinpro White Varnish contains an innovative tri-calcium phosphate.Open the unit-dose package of Varnish and dispense the entire content onto the round application guide provided with the packet. Use the applicator brush to thoroughly mix Varnish. Apply Varnish evenly in a thin layer over treatment area(s). For larger surface areas, apply Varnish in sweeping horizontal brush. After application, instruct the patient to close his or her mouth to set the Varnish. No need to use suction. The patient may feel the thin coating when rubbing the treated area with his or her tongue. The treatment period for Varnish is minimally 4 hour.
  Other Names: Fluoride Varnish
  Arms: White Varnish 3M

SUMMARY:
Dental caries is the destruction of the tooth structure in the presence of organic acids produced by cariogenic bacteria located in the dental biofilm (Dowker et al., 1999 and Robinson et al., 2000).Tooth enamel comprises 90% substituted hydroxyapatite (Ca10 (PO4)6(OH) 2), which is subjected to consecutive cycles of demineralization and remineralization. This is an interrupted process, with periods of remineralization and demineralization occurring, depending on the state of the oral environment in terms of the prolonged accumulation and retention of bacterial plaque on the enamel surface (Aoba, 2004).

Oral bacteria ferment carbohydrates to produce organic acids which lower the pH and cause the subsurface dissolution of the hydroxyapatite crystals. Under normal physiological conditions (pH7), saliva is supersaturated with calcium and phosphate ions which diffuse into the vacancies created during acid-mediated demineralization episodes (Dowker et al., 1999 and Robinson et al., 2000). The demineralization of enamel (white spot lesions) is a significant problem during and after orthodontic treatment with prevalence 71.1% and various preventive measures have been suggested to minimize the incidence (Derks et al., 2004 and Al Maaitah et al., 2011).

DETAILED DESCRIPTION:
In orthodontic patients, demineralization usually takes place in the form of white or brown spots on the enamel around the brackets and can lead to cavitation (Al Maaitah et al., 2011). White spot lesions compromise esthetics and can be extremely difficult or even impossible to reverse.

Natural remineralization through saliva involving a mineral gain in the surface layer of white spot lesions has little improvement on the esthetic and structural properties of the deeper lesions (Karlinsey et al., 2009 and Cochrane et al., 2010). Management of white spot lesion should involve methods of both preventing demineralization and encourage the remineralization of existing lesions. In both of these processes, the efficacy of fluoride is well established. Fluoride increases the initial rate of remineralization of early enamel lesions. Consequently, it slows down the caries process and arresting the lesion. Fluoride varnish provides a protective coat over the tooth which adheres longer to the tooth surface (Demito et al., 2004 and Ten Cate et al., 2008).

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging 11-16 years.
2. Good general health.
3. Exhibiting at least 2 white spot lesion in buccal surface of their teeth.

Exclusion Criteria:

1. Chronic use of medication causing dry mouth.
2. Oral ulcer, ulcerous gingivitis, acute bronchial asthma.
3. History of allergic reaction to fluoride or other ingredients in varnish.
4. Refusal of the patient to participate in the trial.
5. Any previous treatment done for white spot lesion.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2017-12-17 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Esthetic effect | 6 months
  Asking patient (yes or No)

SECONDARY OUTCOMES:
Clinical assessment | 6 months
  International Caries Detection and Assessment System (ICDAS II) by score

OTHER OUTCOMES:
Photography | 6 months
  Enamel decalcification index by score

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Al Manyal, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided